CLINICAL TRIAL: NCT02604485
Title: A Single-Dose Open-Label Study of XOMA 358 in Subjects With Congenital Hyperinsulinism (HI)
Brief Title: A Single-Dose Open-Label Study of XOMA 358 in Subjects With Congenital Hyperinsulinism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X358602
Record Dates: First submitted 2015-10-26; First posted 2015-11-13 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Congenital Hyperinsulinism
Keywords: Hypoglycemia; Congenital Hyperinsulinism
MeSH Terms: conditions — Congenital Hyperinsulinism; Hypoglycemia | interventions — KPNA1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Other): XOMA 358 dose level A, dose level B, dose level C, and dose level D.
  Interventions: Drug: Cohort 1; Drug: Cohort 2; Drug: Cohort 3; Drug: Cohort 4

INTERVENTIONS:
Drug: Cohort 1 — XOMA 358 single dose level A administered by an intravenous infusion
Drug: Cohort 2 — XOMA 358 single dose level B administered by an intravenous infusion
Drug: Cohort 3 — XOMA 358 single dose level C administered by an intravenous infusion
Drug: Cohort 4 — XOMA 358 single dose level D administered by an intravenous infusion

SUMMARY:
The purpose of this study is to evaluate the safety and clinical pharmacology of a single dose pharmacokinetics and pharmacodynamics of XOMA 358 in subjects with hypoglycemia associated with congenital hyperinsulinism.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of congenital hyperinsulinism
* Duration of glucose levels less than 70mg/dL, by CGM, for an average of at least 120 minutes a day across baseline Days -3, -2, and -1 with no single duration less than 60 minutes on any of the baseline Days -3, -2, or -1, unless the subject received rescue treatment.
* Can safely washout of background medications used to treat hyperinsulinism.

Exclusion Criteria:

* Use of any agent, such as diazoxide, octreotide, chronic systemic glucocorticoids, or β agonists that may affect glucose metabolism
* Body Mass Index ≥ 35 kg/m2
* Pregnant females, females planning to become pregnant during the course of the study, females who have delivered 3 months before screening, or breastfeeding
* Male subjects who are planning a pregnancy with a female partner during the course of the study or within 4 months after administration of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 42 days
  Safety assessed by treatment-emergent adverse events
Change from baseline in glucose levels as measured using a continuous glucose monitor | 42 days
  Safety assessed by pre- and post-treatment measurements of vital signs and laboratory test results
Fasting and post prandial blood glucose levels | 42 days
  Assessment of blood glucose collected at time points specified in the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Allan Gordon, MD, PhD, Study Director — XOMA (US) LLC
Locations (2):
- Philadelphia, Pennsylvania, United States
- London, United Kingdom